CLINICAL TRIAL: NCT07099703
Title: The Effect of Ahi-Based Education on the Professional Values of Nursing Students: An Experimental Study
Brief Title: Ahi-Based Education on the Professional Values of Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Gamze Saatçi, Research Assistant, Kirsehir Ahi Evran Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025/03/16
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Nursing Students; Professional Values; Education
Keywords: nursing students; professional values

STUDY DESIGN:
Intervention Model Description: Non-randomized intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ahi-Based Education (Experimental): The Ahilik course is based on the Ahilik system. The course covers topics such as morality, etiquette, ethics, values, and professional ethics.
  The Ahilik system offers a noteworthy model in terms of both professional value education and individual ethical development. Ahilik is a guild and craftsmen organization established in Anatolia in the 13th century by Ahi Evran-ı Veli. This system was not only an economic and professional organization but also functioned as a moral, social, and cultural structure. The Ahilik organization aimed not only to impart professional skills to individuals but also to develop behavior based on universal ethical values such as honesty, justice, charity, equality, respect for human rights, and service to society.
  Interventions: Other: Experimental
- Routine education (Active Comparator): Students at Suşehri Health Vocational School in the control group will continue with their current curriculum and will not receive any Ahilik training.
  Interventions: Other: Routine education

INTERVENTIONS:
Other: Experimental — At Kırşehir Ahi Evran University, which is part of the Intervention Group, Ahilik education is a compulsory course within the current curriculum and will be taught over a period of 14 weeks. Ahilik education covers topics such as morality, etiquette, ethics, values, and professional ethics.
  Arms: Ahi-Based Education
Other: Routine education — They will continue with their current curriculum and will not receive any Ahilik training.
  Arms: Routine education

SUMMARY:
In current nursing education programs, professional values education mostly remains at a theoretical level; students' internalization of these values and reflection of them in their behavior is limited. Ahilik is a historical system based on ethical principles, professional responsibility, and a sense of service to society. The aim of this study is to experimentally evaluate the effect of Ahilik-based education on the professional values of nursing students.

Hypotheses H0: There is no significant difference between the professional values of nursing students who receive Ahilik education and those who do not.

H1: The professional values of nursing students who receive Ahilik education are significantly different from those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in the second year of a nursing bachelor's degree program,
* Be willing to participate in the study,
* Be able to actively participate in the training process (no health problems, active student),
* Agree to attend 80% of the designated training sessions.

Exclusion Criteria:

* Those who attend less than 80% of training sessions
* Students who graduated or withdrew before data collection
* Students with a psychiatric diagnosis or health issues that prevent communication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Professional values results | 6 months
  Nurses Professional Values Scale-Revised reflecting the American Nurses Association's code of ethics was developed by Darlene Weis and Mary Jane Schank in 2009 (Weis & Schank, 2009). It was developed to determine the compliance of nurses and nursing students with professional values. The Turkish validity and reliability study of the scale was conducted by Acaroğlu (2014). The 5-point Likert-type scale consists of 26 items. Each item is scored between 5 (most important) and 1 (not important), and these scores are summed to obtain scale scores. Scores that can be obtained from the scale range between 26 and 130. A high score indicates a strong adaptation to professional values. The scale does not include sub-dimensions. In the scale independent of the sub-dimension, there are sub-factors named as caring, professionalism and trust that contribute to the interpretation of the data. The goodness of fit statistics of the scale was found to be at appropriate values, Cronbach's Alpha reliabil

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Korkut, Study Director — TC Erciyes University
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosmai S, Ali J, Allevi D, et al. (2025). The Professional Values of Nursing Students: A Systematic Review. Infermieristica Journal, 4(1), 131-142. http://doi.org/10.36253/if-3539
- [Background] Barsanti JA, Finco DR. Management of post-renal uremia. Vet Clin North Am Small Anim Pract. 1984 May;14(3):609-16. doi: 10.1016/s0195-5616(84)50066-7. No abstract available. PMID 6610983
- [Background] Yüksel, İ. (2019). Ahilik felsefesinden günümüz meslek ahlakı tartışmalarına bir bakış. Bilecik Şeyh Edebali Üniversitesi Sosyal Bilimler Dergisi, 4(2), 500-537.